CLINICAL TRIAL: NCT05068492
Title: A Novel Imaging Based Quantitative Model-aided Detection of Portal Hypertension in Patients With Cirrhosis (CHESS2104): A Prospective, Multicenter Study
Brief Title: A Novel Imaging Based Quantitative Model-aided Detection of Portal Hypertension in Patients With Cirrhosis (CHESS2104)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hepatopancreatobiliary Surgery Institute of Gansu Province (Other)
Collaborators: Portal Hypertension Alliance in China (Unknown)
Responsible Party: Principal Investigator, Xiaolong Qi, Chief, Institute of Portal Hypertension, The First Hospital of Lanzhou University, Hepatopancreatobiliary Surgery Institute of Gansu Province
Other Study IDs: CHESS2104
Record Dates: First submitted 2021-09-27; First posted 2021-10-05 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Portal Hypertension
Keywords: Cirrhosis; Portal hypertension; Artificial intelligence; CT; MRI; Ultrasound
MeSH Terms: conditions — Hypertension, Portal; Fibrosis | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training cohort: Training cohort was set to develop the novel non-invasive model for virtual HVPG
  Interventions: Diagnostic Test: CT; Diagnostic Test: MRI; Diagnostic Test: HVPG; Diagnostic Test: Ultrasound
- Validation cohort: Validation cohort was set to validate the novel non-invasive model for virtual HVPG in different people in same environments
  Interventions: Diagnostic Test: CT; Diagnostic Test: MRI; Diagnostic Test: HVPG; Diagnostic Test: Ultrasound
- Test cohort: Test cohort was set to test the novel non-invasive model for virtual HVPG in different environments
  Interventions: Diagnostic Test: CT; Diagnostic Test: MRI; Diagnostic Test: HVPG; Diagnostic Test: Ultrasound

INTERVENTIONS:
Diagnostic Test: CT — enhanced CT with standard procedure
Diagnostic Test: MRI — enhanced MRI with standard procedure
Diagnostic Test: HVPG — HVPG measurements are performed by well-trained interventional radiologists in accordance with standard operating procedures
Diagnostic Test: Ultrasound — Digestive ultrasound with standard procedure

SUMMARY:
How to construct a novel, non-invasive, accurate, and convenient method to achieve prediction of hepatic venous pressure gradient (HVPG) is an important general problem in the management of portal hypertension in cirrhosis. We plan to investigate the ability of AI analysis of Ultrasound, computed tomography (CT) or magnetic resonance (MR) to establish a risk stratification system and perform tailored management for portal hypertension in cirrhosis.

DETAILED DESCRIPTION:
China suffers the heaviest burden of liver disease in the world. The number of chronic liver disease is more than 400 million. Either viral-related hepatitis, alcoholic hepatitis, or metabolic-related fatty hepatitis, etc. may progress to cirrhosis, which greatly threatens public health. Portal hypertension is a critical risk factor that correlates with clinical prognosis of patients with cirrhosis. According to the Consensus on clinical application of hepatic venous pressure gradient in China (2018), hepatic venous pressure gradient (HVPG) greater than 10,12,16,20 mmHg correspondingly predicts different outcomes of patients with cirrhosis portal hypertension. It is of great significance to establish a risk stratification system and perform tailored management for portal hypertension in cirrhosis. As a universal gold standard for diagnosing and monitoring portal hypertension, HVPG remains limitation for clinical application due to its invasiveness. How to construct a novel, non-invasive, accurate, and convenient method to achieve prediction of HVPG is an important general problem in the management of portal hypertension in cirrhosis.

The development of radiomics technique provides an approach to solve abovementioned clinical issues. Based on artificial intelligence algorithms, radiomics harnesses mineable, high-resolution, and quantitative features from encrypted medical images, along with clinical or genetic data to produce evidence-based decision support system, to achieve the clinical targets including diagnosis, treatment effect evaluation, and prognosis prediction. In this project, aiming at development of a risk stratification system for hypertension management in cirrhosis, we will construct a standard-of-care database and utilize radiomics tool to construct the decision making system. We will take responsibility for achievement of organ and vessel segmentation, radiomic feature selection, and signature construction for prediction of hypertension classification, and accomplish the development of prototype system which would integrate four modules including database management, HVPG risk stratification application module, predicted outcome presentation module, and prognostic information curation module. This project will focus on two aspects which are correspondingly machine learning algorithms optimization and prototype system development, so as to promote the precision medicine in liver disease.

ELIGIBILITY:
Inclusion Criteria:

1. age > 18 years old;
2. confirmed cirrhosis (laboratory, imaging and clinical symptoms);
3. with ultrasound/CT/MRI within 1 month prior to HVPG measurement;
4. written informed consent.

Exclusion Criteria:

1. any previous liver or spleen surgery;
2. liver cancer; chronic acute liver failure;
3. acute portal hypertension;
4. unreliable HVPG or ultrasound/CT/MRI results due to technical reasons.
5. with liver interventional therapy between HVPG and ultrasound/CT/MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Organize paticipating units to collect standard-of-care data including radiological and clinical data. Patients diagnosed with cirrhosis who received HVPG measurement and enhanced abdominal ultrasound/CT/MRI scan should be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-10 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | 24 months
  Accuracy of the novel model for virtual HVPG

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolong Qi, Prof., Principal Investigator — CHESS Center, Institute of Portal Hypertension, The First Hospital of Lanzhou University, Lanzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu Y, Ning Z, Ormeci N, An W, Yu Q, Han K, Huang Y, Liu D, Liu F, Li Z, Ding H, Luo H, Zuo C, Liu C, Wang J, Zhang C, Ji J, Wang W, Wang Z, Wang W, Yuan M, Li L, Zhao Z, Wang G, Li M, Liu Q, Lei J, Liu C, Tang T, Akcalar S, Celebioglu E, Ustuner E, Bilgic S, Ellik Z, Asiller OO, Liu Z, Teng G, Chen Y, Hou J, Li X, He X, Dong J, Tian J, Liang P, Ju S, Zhang Y, Qi X. Deep Convolutional Neural Network-Aided Detection of Portal Hypertension in Patients With Cirrhosis. Clin Gastroenterol Hepatol. 2020 Dec;18(13):2998-3007.e5. doi: 10.1016/j.cgh.2020.03.034. Epub 2020 Mar 21. PMID 32205218
- [Background] Liu F, Ning Z, Liu Y, Liu D, Tian J, Luo H, An W, Huang Y, Zou J, Liu C, Liu C, Wang L, Liu Z, Qi R, Zuo C, Zhang Q, Wang J, Zhao D, Duan Y, Peng B, Qi X, Zhang Y, Yang Y, Hou J, Dong J, Li Z, Ding H, Zhang Y, Qi X. Development and validation of a radiomics signature for clinically significant portal hypertension in cirrhosis (CHESS1701): a prospective multicenter study. EBioMedicine. 2018 Oct;36:151-158. doi: 10.1016/j.ebiom.2018.09.023. Epub 2018 Sep 27. PMID 30268833